CLINICAL TRIAL: NCT03932656
Title: Latent Toxoplasmosis in Females With Borderline Personality Disorder - Occurrence, Clinical Features, and Impact on Effectiveness of Combined Pharmacotherapeutic and Psychotherapeutic Treatment
Brief Title: Latent Toxoplasmosis in Females With Borderline Personality Disorder
Status: Withdrawn | Type: Observational
Why Stopped: Funding issues
Sponsor: Marie Ociskova (Other)
Collaborators: Palacky University (Other); University Hospital Olomouc (Other)
Responsible Party: Sponsor-Investigator, Marie Ociskova, Assistant Professor, Palacky University
Organization: Palacky University (Other)
Other Study IDs: NV19-05-00105
Record Dates: First submitted 2019-04-22; First posted 2019-05-01 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Borderline Personality Disorder; Toxoplasmosis
Keywords: borderline personality disorder; latent toxoplasmosis; Toxoplasma gondii; pharmacotherapy; psychotherapy; clinical features
MeSH Terms: conditions — Borderline Personality Disorder; Toxoplasmosis | interventions — Cognitive Behavioral Therapy; Psychotropic Drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Females with borderline personality disorder
  Interventions: Behavioral: Combined schema-therapy and cognitive behavioral therapy; Drug: Psychopharmaceuticals

INTERVENTIONS:
Behavioral: Combined schema-therapy and cognitive behavioral therapy — A six-week inpatient psychotherapeutic program consisting of one small group and one big group therapy per day, one individual session per week, daily sport activities, imagery and relaxation techniques. The therapeutic approach presents a combination of schema-therapy and cognitive behavioral therapy. Schema-therapy will follow guidelines for the treatment of individuals with borderline personality disorder (Farrell and Shaw 2012). A later step in the therapy - strengthening of the called Healthy Adult (that is the ability to perceive situations realistically, think rationally, plan time, set appropriate goals, or behave assertively) will be done by standard cognitive behavioral strategies (cognitive restructuring, core beliefs work, time planning, problem solving, assertiveness training). A detailed description of the program is going to be published in a paper.
Drug: Psychopharmaceuticals — Pharmacotherapy will be implemented according to the National Institute for Health and Care Excellence guidelines and will target comorbidities if present to such extent that warrants a pharmacological intervention. If not needed, patients will not use medication. Most patients will be recommended to hospitalization by their outpatient psychiatrists who prescribe the medication. If needed, medication will be changed to meet the guideline standards (i.e., tapering off benzodiazepines or augmentation with a mood stabilizer). The medication will be controlled but not directed by the study.

SUMMARY:
Borderline personality disorder is a common mental disorder with core features of affective dysregulation, impulsivity, and identity disturbance. Although this disorder is mostly understood as a result of a combination of biological factors (genes, temperament) and early aversive experiences (often of traumatic nature), recent data suggest that other factors may be important in its development and course. Preliminary findings show that patients with borderline personality disorder have higher prevalence of Toxoplasma seropositivity. This infection may manifest in symptoms such as affective dysregulation, aggression, suicidality, or anxiousness. As such, it may play a role in the psychopathology of the borderline personality disorder. The aim of this study is to explore the prevalence of Toxoplasma seropositivity in a sample of females with borderline personality disorder, its clinical correlates, and a potential impact on outcomes of an intensive six-week inpatient schema-therapeutic treatment. Results may enrich our understanding of this disorder and lead to improvements of the therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Female
* Borderline personality disorder diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders-5 criteria
* Signed informed consent

Exclusion Criteria:

* Current substance abuse disorder
* Psychotic disorder, bipolar disorder, organic mental disorder current or past
* Severe suicidal risk
* Severe somatic illness (e.g., endocrinopathy, oncologic, hematologic, cardiologic, or neurologic illness)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with borderline personality disorder who will be hospitalized at the psychotherapeutic ward of the university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Immunoglobulin A detection in human serum | 1 day
  ELISA detection of immunoglobulin A specific antibodies - a sensitive and specific marker of acute infection. Index of positivity is higher than 1,1.
Immunoglobulin M detection in human serum | 1 day
  ELISA detection of immunoglobulin M specific antibodies - a highly sensitive marker of acute infection. Index of positivity is higher than 1,1.
Immunoglobulin G detection in human serum | 1 day
  ELISA detection of immunoglobulin G specific antibodies - a marker of undergone infection. The cut-off score for positivity is set at higher than 6,6 IU/ml.
Severity of borderline personality symptoms | 1 year
  Assessed by modified Clinical Global Impression for borderline personality disorder which was developed by Pérez et al (2007). This rating scale measures severity of the nine diagnostic criteria of the disorder, along with its overall severity. In each item, a clinician chooses one number of a seven-point scale where 1 = normal, not at all ill and 7 = among the most extremely ill subjects. The scores in the items are not summed. Instead, each of the item enters statistical analyses separately.

SECONDARY OUTCOMES:
Borderline Evaluation of Severity over Time | 1 year
  This self-rating scale evaluates common symptoms of borderline personality disorder during a specified time range (7 days, 30 days, or other) (Pfohl et al. 2009). 15 items divide into three subscales - thoughts and feelings, behaviors (negative), and behaviors (positive). The patient responds to each item on a 5-point scale according to how much the symptom caused her distress, relationship issues, or disability (in the thoughts and feelings and negative behaviors subscales) and how often she engaged in positive behaviors. The total score ranges between 12 and 72, with higher scores indicating more severe symptomatology.
Aggression Questionnaire | 1 year
  The questionnaire, created by Buss and Perry (1992), has 29 items that are divided into four factors - physical aggression, verbal aggression, anger, and hostility. The patient chooses a number from a five-point scale according to how much is each statement characteristic of her. The total score varies from 29 to 145; higher scores indicating more pronounced aggressive tendencies.
Suicide Behaviors Questionnaire-Revised | 1 year
  The questionnaire has four items that evaluate suicidality - a lifetime frequency of suicide ideation and/or attempt, a frequency of suicidal ideation in the last 12 months, a frequency of threats of suicide attempt, and self-reported likelihood of suicidal behavior in the future (Osman et al. 1999). The total score ranges from 3 to 18; higher scores indicate more severe suicidality.
Beck Anxiety Inventory | 1 year
  The self-rating inventory measures 21 symptoms of anxiety in the time span of a week (Beck et al. 1988). The patient evaluates each symptom with a four-point scale where higher scores mean more severe symptomatology. The total score varies from 0 to 63 points.
Beck Depression Inventory-II | 1 year
  The self-rating inventory measures 21 symptoms of depression during the last two weeks (Beck et al. 1996). The patient chooses perceived severity of each symptom. The total score can reach 0 to 63 points, higher scores representing more severe depressive symptomatology.
Dissociative Experiences Scale | 1 year
  The scale focuses on 28 dissociative symptoms that include dissociative amnesia, depersonalization, derealization, and absorption (Bernstein and Putnam 1986). The patient marks a spot on a 10-cm scale according to how often she perceives the symptom. The total score ranges from 0 to 100 - this number denotes how much time the individual spends in dissociative states.
Sheehan Disability Scale | 1 year
  The scale assesses the level of functional impairment in three areas - work/school, social, and family life (Sheehan 1983). The patient chooses a number from 0 to 10 according to how much her mental disorder disrupted her functioning in each area. The total score then ranges from 0 to 30, higher scores meaning larger disability.

OTHER OUTCOMES:
Childhood Trauma Questionnaire | 1 day
  The questionnaire was created by Bernstein et al. (1994) as a screening for history of child abuse and neglect. It consists of 28 items divided into five factors - emotional, sexual, and physical abuse and emotional and physical neglect. In each item, the patient states how often she experienced described situation on a five-point scale (1 = never, 5 = very often). A total score of each subscale is then calculated; higher scores mean more aversive experiences in childhood.
Parental Bonding Instrument Questionnaire | 1 day
  The questionnaire retrospectively evaluates parental attachment (separately for each parent) up to 16 years of age (Parker 1979). It consists of 25 items divided into two subscales - care and overprotection. The patients evaluates each item on a four-point scale according to how much she finds the statement fitting to her parents. The results are separate for the parents. Each of them get two scores - one for care and one for overprotection. The lowest score of the subscales is 0, the highest is 36 (for the care subscale) or 39 points (for the overprotection subscale). The parental bonding then may be assigned into four categories - affectionate constraint, affectionless control, optimal parenting, and neglectful parenting.
Internalized Stigma of Mental Illness Scale | 1 day
  The scale was developed by Ritsher et al. (2003). In 29 items, it measures the extent of internalized stigma (in other words self-stigma). The scale consists of five subscales - alienation, stereotype endorsement, perceived discrimination, social withdrawal, and stigma resistance. Each statement is rated with a four-point scale according to how much the patient agrees with it. The total score lies between 29 and 116 points, higher score indicating more severe self-stigma.
The Experiences in Close Relationship-Revised Questionnaire | 1 day
  The questionnaire evaluates two basic dimensions of adult attachment - attachment-related anxiety and attachment-related avoidance (Fraley et al. 2000). The measurement consists of 36 items, first half assessing the anxiety, the second half evaluating the avoidance. Each item is rated on a seven-point scale according to the level of agreement. There are two resultant scores (one for the anxiety subscale, the other for the avoidance subscale) which present the means of the items in each subscale. These scores can lie between 1 and 7, higher scores indicating more intensive attachment-related anxiety and attachment. By a comparison with norms, it is possible to define four attachment types - secure, dismissing, fearful, and preoccupied.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Ociskova, PhD, Principal Investigator — University Hospital Olomouc, Faculty of Medicine, Palacky University
Locations (1):
- Department of Psychiatry, Palacky University, University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pfohl B, Blum N, St John D, McCormick B, Allen J, Black DW. Reliability and validity of the Borderline Evaluation of Severity Over Time (BEST): a self-rated scale to measure severity and change in persons with borderline personality disorder. J Pers Disord. 2009 Jun;23(3):281-93. doi: 10.1521/pedi.2009.23.3.281. PMID 19538082
- [Background] Perez V, Barrachina J, Soler J, Pascual JC, Campins MJ, Puigdemont D, Alvarez E. The clinical global impression scale for borderline personality disorder patients (CGI-BPD): a scale sensible to detect changes. Actas Esp Psiquiatr. 2007 Jul-Aug;35(4):229-35. PMID 17592784
- [Background] Buss AH, Perry M. The aggression questionnaire. J Pers Soc Psychol. 1992 Sep;63(3):452-9. doi: 10.1037//0022-3514.63.3.452. PMID 1403624
- [Background] Osman A, Bagge CL, Gutierrez PM, Konick LC, Kopper BA, Barrios FX. The Suicidal Behaviors Questionnaire-Revised (SBQ-R): validation with clinical and nonclinical samples. Assessment. 2001 Dec;8(4):443-54. doi: 10.1177/107319110100800409. PMID 11785588
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Bernstein EM, Putnam FW. Development, reliability, and validity of a dissociation scale. J Nerv Ment Dis. 1986 Dec;174(12):727-35. doi: 10.1097/00005053-198612000-00004. PMID 3783140
- [Background] Bernstein DP, Fink L, Handelsman L, Foote J, Lovejoy M, Wenzel K, Sapareto E, Ruggiero J. Initial reliability and validity of a new retrospective measure of child abuse and neglect. Am J Psychiatry. 1994 Aug;151(8):1132-6. doi: 10.1176/ajp.151.8.1132. PMID 8037246
- [Background] Ritsher JB, Otilingam PG, Grajales M. Internalized stigma of mental illness: psychometric properties of a new measure. Psychiatry Res. 2003 Nov 1;121(1):31-49. doi: 10.1016/j.psychres.2003.08.008. PMID 14572622
- [Background] Parker G, Tupling H, Brown LB. A Parental Bonding Instrument. British Journal of Medical Psychology 52: 1-10, 1979.
- [Background] Brennan KA, Clark CL, Shaver PR. Self-report measurement of adult attachment: An integrative overview. In Simpson JA & Rholes WS (Eds.), Attachment theory and close relationships (pp. 46-76). New York: Guilford Press; 1998.
- [Background] Fraley RC, Waller NG, Brennan KA. An item response theory analysis of self-report measures of adult attachment. J Pers Soc Psychol. 2000 Feb;78(2):350-65. doi: 10.1037//0022-3514.78.2.350. PMID 10707340
- [Background] Sheehan DV. The Anxiety Disease. New York: Scribner's; 1983.
- [Background] Farrell JM, Shaw IA. Group schema therapy for borderline personality disorder: A step-by-step treatment manual with patient workbook. First edition. Chichester, United Kingdom: John Wiley & Sons Ltd; 2012.